CLINICAL TRIAL: NCT04170660
Title: AngioCHIC : Interest of sFlt1/PlGF Ratio at Obstetric Emergencies
Brief Title: Interest of sFlt1/PlGF Ratio at Obstetric Emergencies
Acronym: AngioCHIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: AngioCHIC
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Suspected Placental Dysfunction, Ruled Out; Pregnancy Complications; Pre-Eclampsia
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic test — During a vascular check-up usually prescribed, an additional blood sample is taken to allow the determination of the sFlt1/PlGf ratio.

SUMMARY:
In patients with suspected placental vascular disease who do not require hospitalization, the use of the sFlt-1 (Soluble FMS like tyrosin-kinase-1)/PlGF (Placental Growth Factor)/ assay can most likely help teams to define the best possible management.

DETAILED DESCRIPTION:
Preeclampsia is a serious obstetric condition, affecting 2 to 5% of pregnancies and associated with maternal hypertension and renal dysfunction. It is a constant concern of obstetrical teams in the pre and post partum period. In case of diagnosis in the emergency unit, patients are usually hospitalized. However, in the case of a diagnosis of preeclampsia has been invalidated, but in presence of isolated or frustrated clinical functional signs, in the case of a history of placental vascular pathology, obstetric teams implement surveillance strategies that are binding on the patients.

The sFlt-1/ PlGF assay has a high negative predictive value for the coming week.

The use in clinical practice of these two biomarkers in the indication of negative prediction at one week could help teams in their management but the interest of this use needs to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Pregnant patients term ≥ at 24 weeks of amenorrhoea (SA),
* Management in obstetrical emergencies and at the Centre Hopsitalier Intercommunal (CHI) de Créteil functional exploration center, with prescription of a vascular-renal check-up (BVR) ((proteinuria/creatinuria ratio, blood count, platelets, blood ionogram, creatinemia, transaminases (ASAT, ALAT), haptoglobulinemia, lactate dehydrogenase (LDH), TP).
* Presenting either one of the following isolated or associated clinical parameters:
* HyperTension
* urinary tape proteinuria
* functional signs of hypertension (headaches, phosphenes, accouphènes)
* live osteotendinous reflexes
* epigastric pains
* weight gain, lower limb edema, facial edema
* oliguria
* vomiting
* or one of the following isolated or associated ultrasound parameters:
* fetal hypotrophy, fetal growth deflection
* fetal Doppler abnormalities (umbilical Doppler, cerebral Doppler)
* ooligo-anamnios with intact membranes
* patient who has been informed and has given her oral non-opposition

Exclusion Criteria:

* Diagnosis of preeclampsia
* Refusal of the patient
* Patient whose symptomatology (clinical or paraclinical) leads to a decision to be hospitalized
* Age < 18 years old
* Non-affiliation to the general social security system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women suspected of placental vascular disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reconvening period in patients with an sFlt1 (Soluble FMS like tyrosin-kinase-1)/PlGF (Placental Growth Factor) ratio <38 (day) | trough participation period, an average of 4 months
  At the end of pregnancy, calculation of the average time between the 1st consultation and the 1st reconvening in patients with an sFlt1/PlGF ratio <38, unknown during pregnancy, to determine if consultations could have been avoided.

SECONDARY OUTCOMES:
reconvening period in patients with an sFlt1/PlGF ratio between 38 and 85 (day) | trough participation period, an average of 4 months
  rate of reconvening
reconvening period in patients with an sFlt1/PlGF ratio superior to 85 (day) | trough participation period, an average of 4 months
  rate of reconvening
blood pressure (mmHg) | trough participation period, an average of 4 months
  Blood pressure higher than 140/90 mm Hg
number of patients with functional signs of hypertension | trough participation period, an average of 4 months
  phosphenes, accouphens, headaches, epigastric bar, edema
number of patient with abnormal vascular and renal blood tests | trough participation period, an average of 4 months
  platelets, transaminase, uric acid, ionogram
proteinuria (mg/mmol) | trough participation period, an average of 4 months
  urine protein-creatinine (P/C) ratio, mg/mmol
Intra Uterine growth restriction (IUGR) | trough participation period, an average of 4 months
  estimate foetal weight < 10 percentile or < 5 percentile
fetal echography | trough participation period, an average of 4 months
  umbilical and/or cerebral doppler
term of delivery (weeks of gestation) | at birth
  Analysis of term delivery with stratification by sFlt-1/PlGF ratio
fetal weight at birth (g) | at birth
  Analysis of fetal weight with stratification by sFlt-1/PlGF ratio
number of hospitalized new born | at birth
  Analysis of number of hospitalized new born with stratification by sFlt-1/PlGF ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No